CLINICAL TRIAL: NCT04092309
Title: Effect of Angiotensin Converting Enzyme and Sacubitril Valsartan in Left Atrial and Left Ventricular Performance, as Assessed With 3D Echocardiography, in Patients After Bone Marrow Transplantation.
Brief Title: Effect of Angiotensin Converting Enzyme and Sacubitril Valsartan in Patients After Bone Marrow Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Principal Investigator, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACE_SAVA_3Decho_BMT
Record Dates: First submitted 2019-09-14; First posted 2019-09-17 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Hematopoietic Stem Cell Transplantation; Cardiotoxicity
Keywords: Cardio-oncology
MeSH Terms: conditions — Cardiotoxicity | interventions — Angiotensin-Converting Enzyme Inhibitors; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: one group after bone marrow transpalntation treated with ACE one group after bone marrow transpalntation treated with sacubitril-valsartan one group after bone marrow transpalntation treated with none of these (control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACE group (Other): patients after bone marrow transplantation will be treated with ACE inhibitor
  Interventions: Drug: ACE inhibitor, Sacubitril-Valsartan
- Sacubitril Valsartan group (Other): patients after bone marrow transplantation will be treated with sacubitril valsartan
  Interventions: Drug: ACE inhibitor, Sacubitril-Valsartan
- Control group (Other): patients after bone marrow transplantation will be treated neither with ACE i nor with sacubitril valsartan
  Interventions: Drug: ACE inhibitor, Sacubitril-Valsartan

INTERVENTIONS:
Drug: ACE inhibitor, Sacubitril-Valsartan — Search for Protective effect after chemotherapy and bone marrow transplantation
  Other Names: Sacubitril-Valsartan

SUMMARY:
The purpose of the present study is to investigate the effect of ACE inhibitors and the sacubitril-valsartan complex in bone marrow transplant patients by assessing cardiovascular and endothelial parameters in order to search for a potent protective role.

DETAILED DESCRIPTION:
The purpose of the present study is to investigate the effect of ACE inhibitors and the sacubitril-valsartan complex in bone marrow transplant patients in preventing cardiotoxicity when administered immediately after transplantation.

The effect of medication will be studied in detail:

i) in global longitudinal strain of left ventricle (GLS), ii) in the volume change of the right and the left ventricle, through the cardiac cycle using 3D echocardiography, iii) in the Myocardial Work Index (MWI) of the left ventricle, with a strain -pressure curve study iv) in the 4D strain of the left atrium, v) in elastic properties of aorta (pulse wave velocity (PWV), central systolic pressure (CSBP-mmHg) and augmentation index (Aix%), vii) in permeability of glycocalyx and viii) in serum biomarker values, namely troponin I high sensitivity and atrial natriuretic peptide (NT-proBNP).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents male and female
* that have just been treated with bone marrow transplantation due to haematological malignancies.

Exclusion Criteria:

* Coronary Artery Disease
* Permanent Atrial Fibrilation
* Signs of Left Ventricular Hypertrophy on electrocardiography or echocardiography
* Left ventricle Ejection Fraction<50% or segmental wall motion abnormalities of left ventricle
* More than moderate valvular disease
* Primary Myocardiopathy
* Blood Pressure<90 mmHg
* GFR<30 ml/min/1,73m2
* Unwilling to recruit
* Uncontrolled Arterial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Effect of treatment in Left Ventricular Function | 2 years
  Left Ventricular Function is assessed by calculating Ejection fraction by 3D echocardiography.
Effect of treatment in left ventricular function | 2 years
  Left Ventricular function is assessed by Global Longitudinal Strain by speckle tracking echocardiography
Effect of treatment in arterial stiffness | 2 years
  Arterial Stiffness is evaluated by Pulse Wave Velocity
Effect of treatment in glycocalyx thickness | 2 years
  Glycocalyx thickness is assessed by measuring perfused boundary region (PBR) of the sublingual arterial microvessels (range 5-25 µm

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, Assoc. Prof, Principal Investigator — Athens University
Locations (1):
- "Attikon" University General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katogiannis K, Ikonomidis I, Farmakis D, Thymis J, Stamouli M, Koliou GA, Makavos G, Tsilivarakis D, Vythoulkas D, Tsirigotis P. Effect of Sacubitril/Valsartan or Enalapril on Left Ventricular Function in Patients With Hematologic Malignancies Treated With Bone Marrow Transplantation: A Randomized Controlled Trial. JACC Adv. 2025 Mar;4(3):101628. doi: 10.1016/j.jacadv.2025.101628. Epub 2025 Feb 20. PMID 39983618